CLINICAL TRIAL: NCT07057583
Title: A Pilot Study of 13Carbon-Based Deep Labeling of Bone Marrow Cells to Map Their Utilization of Extracellular Metabolites
Brief Title: A Study of Carbon 13-based Deep Labelling of Bone Marrow Cells
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-003478; NCI-2025-01095 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-003478 (Other: Mayo Clinic in Rochester); HT9425-24-1-0619 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance (MGUS); Non-IgM Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Group I: Patients undergo blood collection and bone marrow aspiration as part of their standard care and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Observational Group II: Healthy volunteers undergo blood collection and bone marrow aspiration on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates a novel laboratory method to study how certain bone marrow cells in the body take up nutrients from their environment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate differences in the amount of extracellular uptake of glucose and amino acids (AAs) between pre-malignant clonal plasma cells (cPCs) and polyclonal plasma cells (pPCs).

OUTLINE: This is an observational study. Participants are assigned to 1 of 2 groups.

GROUP I: Patients undergo blood collection and bone marrow aspiration as part of their standard care and have their medical records reviewed on study.

GROUP II: Healthy volunteers undergo blood collection and bone marrow aspiration on study.

ELIGIBILITY:
Inclusion Criteria:

* All Participants:

  * At least age 18 years or older
  * Able to provide informed consent
* MGUS Cohort:

  * International Myeloma Working Group (IMWG) criteria for the diagnosis of non-IgM MGUS

Exclusion Criteria:

* All Participants:

  * Unable to provide consent
  * Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) >1
  * Prior history of adverse events with conscious sedation
  * Ongoing use of immunosuppressive medications
  * All known pregnant and lactating women will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of monoclonal gammopathy of undetermined significance (MGUS) and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Extracellular uptake of glucose and amino acids (AAs) between pre-malignant clonal plasma cells (cPCs) and polyclonal plasma cells (pPCs) | Up to 30 days
  Assessed by evaluating blood and bone marrow aspirate samples for mean 13Carbon (13C) percentage enrichment of the mass isotopomers of interest of at least 6 (i.e. the difference between a mean 13C percentage enrichment of a particular mass isotopomer is 12% in the MGUS group and 6% in the healthy participant group or vice versa) using a 2-group t-test with a 2-sided significance level of 0.01.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson I. Gonsalves, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials